CLINICAL TRIAL: NCT00653094
Title: An Open Label, Prospective, One Arm, Feasibility, Study for The Use of Halevy Kit for the Treatment of Perianal Fistulas in Patients With Crohn's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ResQ Medical Ltd (Other)
Responsible Party: Elisha Yalin, ResQ Medical Ltd
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H.K.prot.02-03-08
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2008-04-04 (Estimated); Status verified 2008-04

CONDITIONS: Crohn Disease; Fistula
Keywords: crohn; fistula; surgery; fibrin glue; seton drainage
MeSH Terms: conditions — Crohn Disease; Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Other)
  Interventions: Device: Halevy kit

INTERVENTIONS:
Device: Halevy kit — the use of Halevy kit in Crohn patients with Fistulas

SUMMARY:
Today, there is no available equipment specifically designed for the procedure of instillation of fibrin glue for the repair of perianal fistulae. The currently used equipment involves surgical tools generally used for fistula surgeries, and injection syringes designed for general use. The injection of biological adhesives is performed using standard adhesive syringes that are not specially designed for use in perianal fistulae. The use of the semi-flexible metal probes can cause trauma to tissue and injure the fistula tract, creating an additional path, and the injection syringe and catheter are often inconvenient for perianal use. This study was design to test the use of Halevy kit, by gastroenterology specialist, as a non traumatic probing, mechanical debridement and injecting or inserting device for treatment substances in perianal fistulas. In this study a gastroenterologist will perform the procedure, in each procedure a trained colorectal surgeon will be present during the surgery to oversee the procedure and to provide surgical help if required.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female age greater than 18
* Patients suffering from Crohn's disease
* Patients with any number of simple or complex fistulas who require surgical intervention, requiring the insertion of a drain (Seton) into the fistula tract, and/or injection of biologic adhesive, or an anal fistula plug
* Able and willing to sign an informed consent
* Patient will be available for follow up.

Exclusion Criteria:

* Pregnant or lactating woman. Woman of childbearing potential will undergo a pregnancy test at the beginning of the trial
* Known immunodeficiency.
* Exclusion Criteria for injecting biologic adhesive:

  * Known allergy to fibrin glue or one of its components.
  * An undrained perianal abscess, diagnosed by a physical examination or imaging methods.
* Known Alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-06 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Success of cannulation of the perianal fistula using the Pathway Probe Catheter will be evaluated | after sugery
Success in using the cleaning brush in preparing the fistula for biologic adhesive injection will be evaluated | after surgery
Success in inserting a draining Seton into the fistula tract by the Halevy kit | after surgery
Success of injecting biologic adhesive into the fistula tract using the designated catheter will be evaluated | after surgery

SECONDARY OUTCOMES:
Control of sphincter will be evaluated by -the Cleveland continence score | after follow up
Discharge from fistula will be evaluated by a questionnaire comparing the situation before and after surgery. | after follow up
Healing of the fistula will be evaluated by a physical examination | after follow up

CONTACTS AND LOCATIONS:
Overall Officials: Eran MR Goldin, Prof, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah medical center, Jerusalem, Israel